CLINICAL TRIAL: NCT06404658
Title: Analgesic Efficacy of Genicular Nerve Block Versus Local Anaesthetic Infiltration Between Popliteal Artery and Capsule of the Knee (IPACK Block ) in Patients Undergoing Anterior Cruciate Ligament (ACL) Repair by Knee Arthroscopy . A Randomized Controlled Prospective Study .
Brief Title: Analgesic Efficacy of Genicular Nerve Block Versus (IPack Block ) in Patients Undergoing (ACL) Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mariana Soliman, Lecturer of anaesthesia, surgical intensive care and pain managment, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMBSUREC/02012024/Kamal
Record Dates: First submitted 2024-04-08; First posted 2024-05-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): did not receive any block just spinal anathesia.
- Genicular nerve block (Active Comparator): patients who receive Genicular nerve block with spinal anathesia .
  Interventions: Procedure: Genicular nerve block
- IPACK block (Active Comparator): patients who receive IPACK block with spinal anathesia.
  Interventions: Procedure: Genicular nerve block

INTERVENTIONS:
Procedure: Genicular nerve block — patients who receive Genicular nerve block with spinal anathesia .
  Arms: Genicular nerve block; IPACK block

SUMMARY:
One of the most common injuries to the knee is an anterior cruciate ligament (ACL) sprain or tear due to trauma ACL damage is crippling and often requires repair with an arthroscopic method, which is an outpatient surgery. Nevertheless, patients experience severe postoperative pain on the first day after the ACL reconstruction.Efficient postsurgery pain management is an important part of patient recovery that is also crucial for their satisfaction.

DETAILED DESCRIPTION:
The optimum role of peripheral nerve blocks in ACL reconstruction continue to be debated as a component of multi-modal analgesia . As such ,an ideal block for ACLR would target sensation but not motor function,have minimal complication risk,and be easily reproducible The genicular nerves include branches from the femoral, common peroneal, saphenous, tibial, and obturator nerves which innervate the knee capsule . The superolateral, superomedial, and inferomedial On the other hand, the interspace between the Popliteal Artery and Capsule of the Knee (IPACK) block provides analgesia on the posterior knee joint, and the application of a genicular or IPACK block has been be associated with promising outcomes following the ACLR surgery

ELIGIBILITY:
Inclusion Criteria:

- Patient age from 18 to 45 years old Patient status ASA I - II Patient body mass index (BMI) <40 kg/m2

Exclusion Criteria:

* -Patients were excluded if they refused consent.
* Patients who are Not cooperative.
* BMI >40 kg/m2.
* Allergy to local anesthetics.
* Patients with anticoagulation or bleeding problems.
* Previous nerve dysfunction.
* Physical status ASA class IV.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
VAS score | 48 hour
  Measuring pain intensity regarding mean visual analogue score (VAS score ) ranging from 0 (no pain) to 10 (the worst imaginable pain.

SECONDARY OUTCOMES:
Ambulatory score | Within 48 hour
  Ambulatory score from ( 0 to 2) (score of 0) is assigned if the activity cannot be performed despite substantial help
  (score of 1 )is assigned if the activity is performed using personal physical support.
  (score of 2) is assigned if the activity is performed independently.
Time of first rescue analgesia | within 24 hour
  the time to ask for the first post operative analgesia
Total opioid consumption post operative | Within 24 hour
  Total opioid consumption post operative
Incidence of occurrence of systemic toxicity | Within 24 hour
  ( hypotension ,arrthymias, bradycardia, cardiac arrest, oral numbness and convulsions
The length of hospital stay . | within one week
  The length of hospital stay .

CONTACTS AND LOCATIONS:
Locations (1):
- Benisuef University Hospital, Benisuef, Egypt